CLINICAL TRIAL: NCT02042235
Title: Parent-implemented Intervention for Very Preterm Children With Language Delay
Brief Title: Very Preterm Children With Language Delay and Parent Intervention
Acronym: EPILANG
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: difficulted recruiting
Sponsor: Lille Catholic University (Other)
Collaborators: Ministry of Health, France (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RC-P0027
Record Dates: First submitted 2014-01-20; First posted 2014-01-22 (Estimated); Last update posted 2020-03-03 (Actual); Status verified 2020-03

CONDITIONS: Preterm Birth; Language Development; Speech Therapy
Keywords: prematurity; language; parent-implemented intervention; speech therapy; neurodevelopment
MeSH Terms: conditions — Premature Birth; Communication Disorders; Language

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Parent-implemented language intervention (Experimental): In the intervention group, the techniques and attitudes favouring use of oral language will be taught to the parents during 15 sessions with the parent(s) and child.
  Interventions: Behavioral: Parent-implemented intervention
- Control group (No Intervention): The control group will benefit from the actual routine care for children with language delay before the age of 3 years. In order to provide them the best routine care, the psychologist will provide some advice to the parents to enhance their child's language (e.g.: using life situations to talk with the child and encourage him/her to talk …).

INTERVENTIONS:
Behavioral: Parent-implemented intervention — In order to achieve the programme of parent-implemented language intervention, a detailed protocol for speech therapists recruited and trained for the present study has been established. The techniques and attitudes favouring use of oral language will be taught to the parents during 15 sessions with the parent(s) and child.
  Arms: Parent-implemented language intervention

SUMMARY:
In studies of children born at term, language delay at the age of 2 years exhibits a spontaneously favourable course in 30 to 50% by the age of 3 years. In France, there is no recommendation for speech therapy before the age of 3 years. However, for term-born children, parent-implemented language interventions conducted during the third year of life have already shown a positive short-term effect on language skills. In these interventions, a skilled interventionist, generally a speech therapist, teaches parents how to use specific language strategies with their child.

The investigators' hypothesis is that such parent-implemented interventions would be particularly appropriate at short and medium term for the improvement of linguistic performances in very preterm children, a population with a high prevalence of early language delay. Currently, there is an opportunity to partly nest an intervention trial in a national prospective population-based cohort of very preterm children, the EPIPAGE (Etude EPIdémiologique sur les Petits Ages GEstationnels) 2 cohort, which has included 5 000 babies born alive in France in 2011. This situation provides considerable methodological advantages.

DETAILED DESCRIPTION:
EPILANG is an open randomized controlled study, in which the final assessment of the children (endpoint) will be conducted by professionals blinded to the treatment group.

Some eligible children will first be screened using the parental questionnaire at 24 months corrected age (CA) of the EPIPAGE 2 cohort. Children with language delay, defined as no words combination and/or less than 30 words from Mac Arthur CDI - short version, and free of exclusion criteria, will be invited to an inclusion visit at 30 months CA, if they are in an EPIPAGE 2 centre participating in the EPILANG trial.

During the inclusion visit, inclusion criteria and the absence of exclusion criteria will be checked, data useful for the study will be collected, and the informed consent of the parents collected. The child will then be randomized either in the control or the intervention group if language delay is still present, defined by a score < 10th percentile at the Mac Arthur CDI. Twins, if both included, will be included in the same group, otherwise only the twin with a language delay will be randomized.

The intervention is organized in 15 weekly one-hour sessions with the child, one or both parents and a speech therapist recruited and trained for the study. Maximum duration for the intervention will be 6 months per child, because some sessions can be missed or delayed. Parents' participation will be recorded.

The usual "wait-and-see" attitude will be provided to the control group, together with basic advice to enhance the child's language at home.

In both groups, audition will be checked by an otolaryngology specialist, following professional recommendations, and care will be provided in case of hearing deficit, if appropriate.

At 3 years CA, a neuropsychological evaluation will be performed by trained psychologists for both groups, blinded for the allocation group. Behaviour will be evaluated with a validated parental questionnaire.

The analysis will be according to intention to treat.

ELIGIBILITY:
Inclusion Criteria:

* Child born at 24 to 31+6 weeks' gestation, whose parents did not refuse collection of follow-up data
* Child aged 30 ± 2 months corrected age (CA) at inclusion
* Child with language delay at 24 months CA, defined as the absence of word combination and/or expressive vocabulary of less than 30 words according to the short version of the French Mac Arthur Communication Developmental Inventories (CDI), whose language delay is confirmed at 30 months CA i.e. without word combination and/or an expressive vocabulary below the 10th percentile on the French CDI.
* Child with a global Developmental Quotient (DQ) ≥ 55 at 30 months CA
* Child whose parents accept participation in this study
* Child with French health insurance coverage

Exclusion Criteria:

* Child with neurological sequelae (delay or disability) and who is unable to walk without assistance at 24 months CA or who has a global DQ < 55 on the revised Brunet-Lézine (BLR) scale at 30 months CA.
* Blindness
* Deafness defined by the prescription of a hearing aid
* Child with a chromosomal or other condition that could interfere with language development
* Parents who do not speak French at all
* Triplets

Ages: 28 Months to 32 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 67 (Actual)
Dates: Start 2014-01; Primary Completion 2018-01-31 (Actual); Study Completion 2018-01-31 (Actual)

PRIMARY OUTCOMES:
language score of the Developmental Neuropsychological assessment (NEPSY) | at 36 months of corrected age
  For the main outcome, mean language score on the NEPSY at the final visit, our primary endpoint, will be compared between groups using linear regression

SECONDARY OUTCOMES:
Other scores of the NEPSY battery | at 36 months of corrected age
  To evaluate the child's neuropsychological functioning
Strengths and Difficulties Questionnaire | at 36 months of corrected age
Parenting Stress Index (PSI) questionnaire | at 36 months of corrected age

CONTACTS AND LOCATIONS:
Overall Officials: Amélie Lansiaux, MD, PhD, Study Chair — Groupment des Hôpitaux de l'Institut Catholique de Lille; Marie-Laure Charkaluk, MD, PhD, Study Director — Hôpital Saint-Vincent-de-Paul, GHICL
Locations (15):
- France (15):
  - Centre Hospitalier, Arras
  - Centre Hospitalier Universitaire, Caen
  - Centre Hospitalier Universitaire, Lille
  - Hôpital Saint Vincent de Paul (GHICL), Lille
  - Hôpital femme mère enfant, Lyon
  - Centre Hospitalier Universitaire, Marseille
  - Centre Hospitalier Universitaire, Nantes
  - AP-HP Hôpital Antoine Béclère, Paris
  - Hôpital Necker, Paris
  - HôpitalCochin - Port Royal, Paris
  - Centre Hospitalier, Roubaix
  - Centre hospitalier Universitaire, Rouen
  - Centre Hospitalier Universitaire, Strasbourg
  - Centre Hospitalier Universitaire, Tours
  - Centre Hospitalier, Valenciennes